CLINICAL TRIAL: NCT03157167
Title: An Evaluation of the Safety of Escalating Doses of Tc 99m Tilmanocept by Intravenous (IV) Injection and a Comparison to Subcutaneous (SC) Injection in Human Immunodeficiency Virus (HIV) Subjects Diagnosed With Kaposi Sarcoma (KS)
Brief Title: An Evaluation of Tc 99m Tilmanocept by Intravenous (IV) and Subcutaneous (SC) Injection in Kaposi Sarcoma (KS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Navidea Biopharmaceuticals (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: NAV3-24; 1R44CA192859-01 (NIH)
Record Dates: First submitted 2017-05-04; First posted 2017-05-17 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2020-07

CONDITIONS: Kaposi Sarcoma; HIV Infections
Keywords: Kaposi Sarcoma, KS, HIV
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections | interventions — technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 100 mcg/5 mCi Tc99m-Tilmanocept (Experimental): Four subjects will receive a single IV injection of 100 micrograms of Tc99m tilmanocept radiolabeled with 5 mCi.
  Interventions: Drug: Tc99m-tilmanocept
- 100 mcg/10 mCi Tc99m-Tilmanocept (Experimental): Four subjects will receive a single IV injection of 100 micrograms of Tc99m tilmanocept radiolabeled with 10 mCi.
  Interventions: Drug: Tc99m-tilmanocept
- 200 mcg/5 mCi Tc99m-Tilmanocept (Experimental): Up to six subjects will receive a single subcutaneous injection and a single IV injection of 200 micrograms of Tc99m tilmanocept radiolabeled with 5 mCi.
  Interventions: Drug: Tc99m-tilmanocept

INTERVENTIONS:
Drug: Tc99m-tilmanocept — Tilmanocept is a radiotracer that accumulates in macrophages by binding to a mannose binding receptor that resides on the surface.
  Other Names: Lymphoseek

SUMMARY:
To determine the safety of escalating IV doses of Tc 99m tilmanocept in HIV (human immunodeficiency virus) subjects with confirmed KS and to compare results obtained from subcutaneous and IV administrations of Tc 99m tilmanocept in the same subjects.

DETAILED DESCRIPTION:
This is a Manocept Platform prospective, single-center, open-label, non-randomized, dose escalation, comparative, safety study of intravenously and subcutaneously injected Tc 99m tilmanocept in the localization and detection of cutaneous and non-cutaneous KS tumor(s) in subjects with biopsy-confirmed KS. Three IV doses (µg/mCi) of tilmanocept will be evaluated in three cohort groups. One subcutaneous dose will be evaluated in cohort group 3.

This study is designed to evaluate the safety and tolerability of escalating doses of IV Tc 99m tilmanocept and to compare results obtained from IV and subcutaneous administrations of Tc 99m tilmanocept in the same subjects. Whole body planar as well as SPECT/CT imaging will be performed to provide greater resolution of areas of Tc 99m tilmanocept localization. A biopsy of a non-visceral KS lesion will be taken to correlate pathology with Tc 99m tilmanocept localization.

This study is designed to evaluate the use of Tc 99m tilmanocept as an imaging agent in HIV-positive subjects with known KS by evaluating localization in known and unknown cutaneous and non-cutaneous lesions.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has provided written informed consent with HIPAA authorization before the initiation of any study-related procedures.
2. The subject is at least 18 years of age at the time of consent.
3. The subject is HIV positive.
4. The subject has a biopsy-confirmed diagnosis of KS and is classified into one of the categories below:

   1. Confirmed cutaneous KS/oral lesions without edema.
   2. Confirmed cutaneous KS/oral lesions with edema.
   3. Confirmed cutaneous KS/oral lesions with or without edema and suspected non-cutaneous KS due to clinical symptomology or confirmed non-cutaneous KS lesion(s).

Exclusion Criteria:

1. The subject is pregnant or lactating.
2. The subject has received chemotherapy or radiation therapy to KS sites within six weeks of enrollment.
3. The subject has known sensitivity to dextran.
4. The subject has received an investigational product within 30 days prior to the Tc 99m tilmanocept administration on Day 1.
5. The subject has received any radiopharmaceutical within 7 days prior to the administration of Tc 99m tilmanocept on Day 1.
6. Any condition that, in the clinical judgment of the treating physician, is likely to prevent the subject from complying with any aspect of the protocol or that may put the subject at unacceptable risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Blue, MD, Study Director — Navidea Biopharmaceuticals
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cope, F.O., W. Metz, et al. Innovations in receptor-targeted precision imaging at Navidea: diagnosis up close and personal. Nature Outlook (31 October 2013); S125-S129.
- [Result] Cope FO, Abbruzzese B, Sanders J, Metz W, Sturms K, Ralph D, Blue M, Zhang J, Bracci P, Bshara W, Behr S, Maurer T, Williams K, Walker J, Beverly A, Blay B, Damughatla A, Larsen M, Mountain C, Neylon E, Parcel K, Raghuraman K, Ricks K, Rose L, Sivakumar A, Streck N, Wang B, Wasco C, Williams A, Schlesinger LS, Azad A, Rajaram MVS, Jarjour W, Young N, Rosol T, McGrath M. Corrigendum to the inextricable axis of targeted diagnostic imaging and therapy: An immunological natural history approach [Nucl Med Biol 43 (2016) 215-225]. Nucl Med Biol. 2016 Dec;43(12):837. doi: 10.1016/j.nucmedbio.2016.10.001. No abstract available. PMID 27866590

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject was enrolled and injected with Tc 99m tilmanocept but after experiencing an AE (anxiety) did not undergo imaging and withdrew from the trial.
  The safety population is defined as any subject that was injected with Tc 99m tilmanocept (15 subjects).
  The intent to diagnose population is defined as all subjects that completed the trial (14 subjects), unless otherwise noted in the outcome measure. One subject in cohort 1 withdrew after injection and was not imaged.
Period: Overall Study
Arm/Group | 100 mcg/5 mCi Tc99m-Tilmanocept | 100 mcg/10 mCi Tc99m-Tilmanocept | 200 mcg/5 mCi Tc99m-Tilmanocept
Started | 5 | 4 | 6
Safety Population | 5 | 4 | 6
Intent to Diagnose Population | 4 (One participant was injected, but they withdrew before imaging could be completed.) | 4 | 6
Completed | 4 | 4 | 6
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 100 mcg/5 mCi Tc99m-Tilmanocept | 100 mcg/10 mCi Tc99m-Tilmanocept | 200 mcg/5 mCi Tc99m-Tilmanocept | Total
Number analyzed (Participants) | 5 | 4 | 6 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 6 | 14
  >=65 years | 1 | 0 | 0 | 1
Age, Continuous [Median (Full Range); unit: years] | 58.0 [45 to 70] | 53.5 [53 to 55] | 38.5 [34 to 67] | 54.0 [34 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 5 | 4 | 6 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 5 | 3 | 5 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 3
  White | 1 | 3 | 3 | 7
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 4 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Safety of Escalating Doses of Tc 99m Tilmanocept in HIV Subjects With Biopsy-confirmed KS.
Description: Cohort 1 (100 mcg/ 5mCi) was conducted first. A safety data review meeting was held after completion of Cohort 1 and again after completion of Cohort 2 at which the principal investigators and sponsor representatives reviewed the safety data to determine whether to proceed to the next cohort. All cohorts were evaluated for safety.
  Safety evaluations included AEs, clinical laboratory tests, vital signs, physical examinations, and ECGs.
  The data table includes the number of safety signals detected during the evaluation for each cohort.
Time Frame: 10 days after IV Tc 99m tilmanocept administration
Population: Safety population, including all subjects injected with Tc99m tilmanocept.
Measure: Number; unit: Safety Signals
Groups:
- 100 mcg/5 mCi Tc99m-Tilmanocept: Four subjects will receive a single IV injection of 100 micrograms of Tc99m tilmanocept radiolabeled with 5 mCi. Note that one additional subject was injected with Tc 99m tilmanocept but withdrew after experiencing anxiety (AE). This brings the safety population for this cohort to 5.
  Tc99m-tilmanocept: Tilmanocept is a radiotracer that accumulates in macrophages by binding to a mannose binding receptor that resides on the surface.
Arm/Group | 100 mcg/5 mCi Tc99m-Tilmanocept | 100 mcg/10 mCi Tc99m-Tilmanocept | 200 mcg/5 mCi Tc99m-Tilmanocept
Number analyzed (Participants) | 5 | 4 | 6
Safety Signals | 0 | 0 | 0

2. Secondary Outcome: Per Subject Localization Rate of Tc 99m Tilmanocept in at Least One KS Suspected or Confirmed Lesion by Planar and/or SPECT/CT Imaging
Description: Presents Tc 99m tilmanocept KS lesion localization in each cohort. IV injections occurred in all three cohorts. SC injections occurred in cohort 3 only.
Time Frame: 10 days after IV Tc 99m tilmanocept administration
Population: The intent to diagnose population, including subjects that were imaged and completed the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | 100 mcg/5 mCi Tc99m-Tilmanocept | 100 mcg/10 mCi Tc99m-Tilmanocept | 200 mcg/5 mCi Tc99m-Tilmanocept
Number analyzed (Participants) | 4 | 4 | 6
Participants
  Localized KS Lesions for IV Injection | 4 | 1 | 0
  Localized KS Lesions for SC Injection: number analyzed (Participants) | 0 | 0 | 6
  Localized KS Lesions for SC Injection | 0 | 0 | 4

3. Secondary Outcome: Qualify and Quantify Tc 99m Tilmanocept Localization Intensity on Imaging With CD206 Locale and Quantity by Histology and IHC in Biopsied KS Lesions to Determine Optimal IV Dose.
Description: Localization intensity for each biopsied and clinically defined lesion was to be determined by Planar and/or SPECT/CT imaging. The results would have been average pixel intensity and percentage above background.
  Note: Cohort 1 was completed before this outcome measure was introduced, therefore no cohort 1 subjects were evaluated for this outcome measure.
Time Frame: 10 days after IV Tc 99m tilmanocept administration
Population: The intent to diagnose population, including subjects that were imaged and completed the trial, excluding cohort 1 as this cohort was completed before this outcome measure was introduced.
Measure: Count of Participants; unit: Participants
Arm/Group | 100 mcg/10 mCi Tc99m-Tilmanocept | 200 mcg/5 mCi Tc99m-Tilmanocept
Number analyzed (Participants) | 4 | 6
Participants
  Subjects Evaluated | 4 | 6
  Biopsy Sample Collection Criteria Met | 0 | 1
  Participants with Valid Biopsy Imaged by SPECT/CT: number analyzed (Participants) | 0 | 1
  Participants with Valid Biopsy Imaged by SPECT/CT |  | 1
  Participants with Valid Biopsy Imaged by Planar Image: number analyzed (Participants) | 0 | 1
  Participants with Valid Biopsy Imaged by Planar Image |  | 0
  Participant with Valid Biopsy that was able to be Quantified: number analyzed (Participants) | 0 | 1
  Participant with Valid Biopsy that was able to be Quantified |  | 0

4. Secondary Outcome: Localization Concordance of Subcutaneous Injection and IV Injection
Description: Per lesion/region concordance of IV vs subcutaneous Tc 99m localization with anatomical areas of active KS defined by confirmed diagnosis or clinical symptomology.
  Note: IV routes of administration are used in all three cohorts. Cohort 3 is the only SC route of administration.
Time Frame: 10 days after IV Tc 99m tilmanocept administration
Population: The intent to diagnose population, including subjects that were imaged and completed the trial.
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | 100 mcg/5 mCi Tc99m-Tilmanocept | 100 mcg/10 mCi Tc99m-Tilmanocept | 200 mcg/5 mCi Tc99m-Tilmanocept
Number analyzed (Participants) | 4 | 4 | 6
Number analyzed (Lesions) | 13 | 9 | 23
Lesions
  Localized Lesions via IV | 3 | 0 | 0
  Localized Lesions via SC: number analyzed (Participants) | 0 | 0 | 6
  Localized Lesions via SC: number analyzed (Lesions) | 0 | 0 | 23
  Localized Lesions via SC |  |  | 1

5. Secondary Outcome: Exploratory: Quantify HHV8 in Biopsied KS Lesions. Mean and Standard Deviation Results.
Description: Quantify HHV8 in biopsied KS lesions by using qPCR. Note: Cohort 1 was completed before this outcome measure was introduced, therefore no cohort 1 subjects were evaluated for this outcome measure.
  If there is identification of HHv8, that would confirm the presence of KS cells in the biopsied tissue.
Time Frame: 10 days after IV Tc 99m tilmanocept administration
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: HHV8 (RFU)
Arm/Group | 100 mcg/10 mCi Tc99m-Tilmanocept | 200 mcg/5 mCi Tc99m-Tilmanocept
Number analyzed (Participants) | 4 | 6
HHV8 (RFU) | 1242.50 (583.635) | 4392.50 (4143.048)

6. Secondary Outcome: Exploratory: Quantify HHV8 in Biopsied KS Lesions. Median Results.
Description: as for outcome 5
Time Frame: 10 days after IV Tc 99m tilmanocept administration
Population: as for outcome 3
Measure: Median (Full Range); unit: HHV8 (RFU)
Arm/Group | 100 mcg/10 mCi Tc99m-Tilmanocept | 200 mcg/5 mCi Tc99m-Tilmanocept
Number analyzed (Participants) | 4 | 6
HHV8 (RFU) | 1171.50 [606.0 to 2021.0] | 4463.50 [73.0 to 10507.0]

ADVERSE EVENTS:
Time Frame: 50 days
Description: No deaths occurred during the trial. No SAEs were reported. No other significant AEs were reported.
Arm/Group | 100 mcg/5 mCi Tc99m-Tilmanocept | 100 mcg/10 mCi Tc99m-Tilmanocept | 200 mcg/5 mCi Tc99m-Tilmanocept
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 1/5 | 1/4 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 mcg/5 mCi Tc99m-Tilmanocept (N=5) | 100 mcg/10 mCi Tc99m-Tilmanocept (N=4) | 200 mcg/5 mCi Tc99m-Tilmanocept (N=6)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Cohort 1 subject who withdrew after injection.
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT03157167/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/67/NCT03157167/SAP_001.pdf
  • Informed Consent Form (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/67/NCT03157167/ICF_002.pdf